CLINICAL TRIAL: NCT04474249
Title: Uppföljning av Patienter Som intensivvårdats för COVID-19
Brief Title: Follow-up of Critical COVID-19 Patients
Acronym: FUP-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EPM-2020-02697
Record Dates: First submitted 2020-06-29; First posted 2020-07-16 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID19; ARDS; AKI; Circulatory Failure; Coagulation Disorder; Inflammatory Response
Keywords: Corona virus; Acute Kidney Injury; SARS; Vasopressor; Respiratory failure
MeSH Terms: conditions — COVID-19; Shock; Hemostatic Disorders; Acute Kidney Injury; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, Whole blood, Dried blood, Serum, EDTA-plasma, Citrate-plasma, cheek swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Patients with PCR-confirmed COVID-19 who were treated in the intensive care unit.

SUMMARY:
The study will follow COVID-19 patients who required intensive care after 3-6 months and one year after discharge from the ICU with functional level as well as organ function to assess recovery after COVID-19. Blood and urine will be collected for biobanking.

DETAILED DESCRIPTION:
The study will follow COVID-19 patients who required intensive care at Uppsala University Hospital and were included in the Uppsala COVID-19 biobank. The patients will be contacted after three to six months for a first follow-up with assessment of functional level in activities of daily life, psychiatric symptoms, neurological symptoms and working capacity as well as specific organ functions. The organ functions will include circulation, respiration, coagulation, immune function and kidney function. In addition, blood and urine will be collected for biobanking.

ELIGIBILITY:
Inclusion Criteria:

* PCR-verified Covid-19
* Treated in ICU

Exclusion Criteria:

* Pregnant of breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | Within 90 days after admission to ICU.
  Death
Mortality | Within 1 year after admission to ICU.
  Death
Renal recovery | At follow-up three to six months after ICU discharge.
  Return of renal function measured as CKD stage.
Renal recovery | At follow-up one year after ICU discharge.
  Return of renal function measured as CKD stage.
Respiratory recovery | Three to six months from discharge from ICU
  Respiratory function as assessed by a clinician
Working capacity | Three to six months from discharge from ICU
  6 min walk test
Quality of life score | Three to six months from discharge from ICU
  Quality of Life assessed using the 36-item short form survey by RAND.
Cognitive recovery | Three to six months from discharge from ICU
  Cognitive screening using the Montreal Cognitive Assessment.
Frailty | Three to six months from discharge from ICU
  Screening for frailty using the Clinical Frailty Scale-9.
Activities of Daily Life | Three to six months from discharge from ICU
  Screening of functional level for Activities of Daily Life using the 5-level EQ-5D.
Anxiety | Three to six months from discharge from ICU
  Screening for anxiety using the Generalised Anxiety Disorder 7-item scale.
Depression | Three to six months from discharge from ICU
  Screening for depression using the Patient Health Questionnaire 9.
Neurological recovery | Three to six months from discharge from ICU
  Neurological function as assessed by a clinician

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on reasonable request.

REFERENCES:
- [Result] E E, R F, Oi E, Im L, M L, S R, E W, C J, M H, A M. Impaired diffusing capacity for carbon monoxide is common in critically ill Covid-19 patients at four months post-discharge. Respir Med. 2021 Jun;182:106394. doi: 10.1016/j.rmed.2021.106394. Epub 2021 Apr 15. PMID 33901787
- [Result] Hultstrom M, Lipcsey M, Wallin E, Larsson IM, Larsson A, Frithiof R. Severe acute kidney injury associated with progression of chronic kidney disease after critical COVID-19. Crit Care. 2021 Jan 25;25(1):37. doi: 10.1186/s13054-021-03461-4. No abstract available. PMID 33494766
- [Derived] Bjarnadottir KJ, Perchiazzi G, Sidenbladh CL, Larina A, Wallin E, Larsson IM, Franzen S, Larsson AO, Sousa MLA, Segelsjo M, Hansen T, Frithiof R, Hultstrom M, Lipcsey M, Pellegrini M. Body mass index is associated with pulmonary gas and blood distribution mismatch in COVID-19 acute respiratory failure. A physiological study. Front Physiol. 2024 Jul 10;15:1399407. doi: 10.3389/fphys.2024.1399407. eCollection 2024. PMID 39050483
- [Derived] Halvorsen P, Hultstrom M, Hastbacka J, Larsson IM, Eklund R, Arnberg FK, Hokkanen L, Frithiof R, Wallin E, Orwelius L, Lipcsey M. Health-related quality of life after surviving intensive care for COVID-19: a prospective multicenter cohort study. Sci Rep. 2023 Oct 21;13(1):18035. doi: 10.1038/s41598-023-45346-2. PMID 37865685
- [Derived] Bark L, Larsson IM, Wallin E, Simren J, Zetterberg H, Lipcsey M, Frithiof R, Rostami E, Hultstrom M. Central nervous system biomarkers GFAp and NfL associate with post-acute cognitive impairment and fatigue following critical COVID-19. Sci Rep. 2023 Aug 12;13(1):13144. doi: 10.1038/s41598-023-39698-y. PMID 37573366
- [Derived] Hultstrom M, Lipcsey M, Morrison DR, Nakanishi T, Butler-Laporte G, Chen Y, Yoshiji S, Forgetta V, Farjoun Y, Wallin E, Larsson IM, Larsson A, Marton A, Titze JM, Nihlen S, Richards JB, Frithiof R. Dehydration is associated with production of organic osmolytes and predicts physical long-term symptoms after COVID-19: a multicenter cohort study. Crit Care. 2022 Oct 21;26(1):322. doi: 10.1186/s13054-022-04203-w. PMID 36271419